CLINICAL TRIAL: NCT04668950
Title: Fluvoxamine for Early Treatment of Covid-19: a Fully-remote, Randomized Placebo Controlled Trial
Brief Title: Fluvoxamine for Early Treatment of Covid-19 (Stop Covid 2)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Covid-19 Early Treatment Fund (Other); McGill University (Other); Cures Within Reach (Other)
Responsible Party: Principal Investigator, Eric Lenze, Principal Investigator, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 202011101
Record Dates: First submitted 2020-12-11; First posted 2020-12-16 (Actual); Results first posted 2022-10-18 (Actual); Last update posted 2022-10-31 (Actual); Status verified 2022-10

CONDITIONS: Covid19; Coronavirus
Keywords: fluvoxamine
MeSH Terms: conditions — COVID-19; Coronavirus Infections | interventions — Fluvoxamine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fluvoxamine (Experimental): Start fluvoxamine 50mg capsule once, then 100mg twice daily. May reduce dose for tolerability reasons. Will be followed in the RCT for approximately 15 days.
  Interventions: Drug: Fluvoxamine
- Placebo (Placebo Comparator): Start placebo one capsule, twice daily. May reduce dose for tolerability reasons. Will be followed in RCT for approximately 15 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fluvoxamine — Up to 200mg per day (2 capsules per day) as tolerated, for approximately 15 days
  Other Names: Luvox
  Arms: Fluvoxamine
Drug: Placebo — Will take 2 capsules per day as tolerated for approximately 15 days
  Arms: Placebo

SUMMARY:
The purpose of this research study is to determine if a drug called fluvoxamine can be used early in the course of the COVID-19 infection to prevent more serious complications like shortness of breath. Fluvoxamine is an anti-depressant drug approved by the FDA for the treatment of obsessive-compulsive disorder. The use of fluvoxamine for the treatment of COVID-19 is considered investigational, which means the US Food and Drug Administration has not approved it for this use.

This study is fully-remote, which means that there is no face-to-face contact; study materials including study drug will be shipped to participants' houses. People around the United States and Canada can participate.

DETAILED DESCRIPTION:
The investigators will randomize approximately 880 participants, age 30 and older, who have tested tested positive for COVID-19 and are currently experiencing mild symptoms. People around the United States and Canada can participate. All interactions for this study will be conducted remotely by videoconferencing, email, or phone.

Screening: All participants will first complete a pre-screen to see if they may be eligible for the study. Once a participant is confirmed eligible and consented, the study team will send the study materials. These materials will consist of study medication and self-monitoring equipment, including an oxygen saturation monitor, blood pressure monitor, and thermometer.

RCT: Participants will be randomly assigned (1:1) to take either fluvoxamine or a placebo. This phase of the study will last approximately 15 days and is double-blinded. Participants will take up to 100mg of fluvoxamine or placebo by mouth twice a day for a daily total of 200mg. Participants will continue this dose for approximately 15 days. Depending on tolerability, the dose may be adjusted. Participants will also complete short 5 minute assessments daily to report the results of self-monitoring (including oxygen level, blood pressure, and temperature), a shortness of breath rating and any adverse events.

Follow-up Phase: The study team will follow participants for approximately 90 days after the end of the randomized phase. If needed, the study team will review medical records to determine the clinical course of participants.

ELIGIBILITY:
Inclusion Criteria:

1. Men and woman age 30 and older;
2. Not currently hospitalized
3. Proven SARS-CoV-2 positive (per lab or physician report).
4. Currently symptomatic with one or more of the following symptoms: fever, cough, myalgia, mild dyspnea, chest pain, diarrhea, nausea, vomiting, anosmia (inability to smell), ageusia (inability to taste), sore throat, nasal congestion.
5. Able to provide informed consent.
6. Upon initial screening, participant reports one of the following risk factors for clinical deterioration: age≥40, racial/ethnic group African-American, Hispanic, or Native American (including more than one race), or 1+ of the following medical conditions which increase risk for developing moderate-severe COVID illness: obesity, hypertension, diabetes, heart disease (coronary artery disease, history of myocardial infarction, or heart failure), lung disease (eg asthma, COPD), immune disorder (eg rheumatoid arthritis, lupus).

Exclusion Criteria:

1. Illness severe enough to require hospitalization or already meeting study's primary endpoint for clinical worsening (eg current O2 saturation <92% on room air, current use of supplemental oxygen to maintain O2 saturation ≥92%).
2. Unstable medical comorbidities (eg decompensated cirrhosis), per patient report and/or medical records.
3. Immunocompromised from the following: solid organ transplant, BMT, high dose steroids (>20mg prednisone per day), or tocilizumab
4. Already enrolled in another COVID 19 medication trial (not including vaccination or prophylaxis trials)
5. Unable to provide informed consent
6. Unable to perform the study procedures
7. Taking donepezil (rationale: donepezil is a S1R agonist), or sertraline (rationale: sertraline is a strong sigma-1 antagonist).
8. Taking warfarin-also known as Coumadin (rationale: increased risk of bleeding), phenytoin (rationale: fluvoxamine inhibits its metabolism), clopidogrel (rationale: fluvoxamine inhibits its metabolism from pro-drug to active drug which raises risk of cardiovascular events), and St John's wort (rationale: fluvoxamine + St John's wort are considered contraindicated because of the risk of serotonin syndrome)
9. Taking SSRIs, SNRIs, or tricyclic antidepressants, unless these are at a low dose such that a study investigator concludes that a clinically significant interaction with fluvoxamine (ie either serotonin syndrome or TCA overdose) is unlikely (examples: participant takes escitalopram but only at 5-10mg daily; that dose plus 200mg fluvoxamine would be insufficient to cause serotonin syndrome; or, participant takes amitriptyline but only at 25mg nightly; even if fluvoxamine inhibits its metabolism, it would be an insufficient dose to cause QTc prolongation or problematic side effects).
10. Individuals who report they have bipolar disorder or are taking medication for bipolar disorder (lithium, valproate, high-dose antipsychotic), unless the investigator concludes that the risk for mania is unlikely (ie it is doubtful that the patient actually has bipolar disorder).
11. Individuals who take alprazolam or diazepam and are unwilling to cut the medication by 25% (rationale: fluvoxamine modestly inhibits the metabolism of these drugs).
12. Participants taking theophylline, tizanidine, clozapine, or olanzapine (drugs with a narrow therapeutic index that are primarily metabolized by CYP 1A2, which is inhibited by fluvoxamine) will be reviewed with a study investigator and excluded unless the investigator concludes that the risk to the participant is low (this would be unlikely; example: participant takes tizanidine only as needed and is willing to avoid it for the 15 days of the study).
13. Received vaccine for COVID-19.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 670 (Actual)
Dates: Start 2020-12-22 (Actual); Primary Completion 2021-09-28 (Actual); Study Completion 2021-09-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (4):
  - Northwestern University, Chicago, Illinois
  - Washington University School of Medicine, St Louis, Missouri
  - University of Utah, Salt Lake City, Utah
  - Fred Hutchinson, Seattle, Washington
- McGill University Health Center, Montreal, Quebec, Canada

REFERENCES:
- [Derived] Reiersen AM, Mattar C, Bender Ignacio RA, Boulware DR, Lee TC, Hess R, Lankowski AJ, McDonald EG, Miller JP, Powderly WG, Pullen MF, Rado JT, Rich MW, Schiffer JT, Schweiger J, Spivak AM, Stevens A, Vigod SN, Agarwal P, Yang L, Yingling M, Gettinger TR, Zorumski CF, Lenze EJ. The STOP COVID 2 Study: Fluvoxamine vs Placebo for Outpatients With Symptomatic COVID-19, a Fully Remote Randomized Controlled Trial. Open Forum Infect Dis. 2023 Aug 8;10(8):ofad419. doi: 10.1093/ofid/ofad419. eCollection 2023 Aug. PMID 37622035

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Fluvoxamine | Placebo
Started | 334 | 336
Completed | 272 | 275
Not Completed | 62 | 61
Not completed — Started medication more than 7 days after symptom onset | 18 | 14
Not completed — Could not confirm started study medication | 15 | 15
Not completed — Could not confirm baseline status | 6 | 2
Not completed — Drop out and did not start medication | 15 | 17
Not completed — Deteriorated at or before baseline assessment | 6 | 9
Not completed — Other | 2 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fluvoxamine | Placebo | Total
Number analyzed (Participants) | 272 | 275 | 547
Age, Customized [Mean (Standard Deviation); unit: years]
  Age | 48 (10.18) | 48 (9.83) | 48 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 169 | 170 | 339
  Male | 103 | 105 | 208
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 35 | 37 | 72
  Not Hispanic or Latino | 234 | 236 | 470
  Unknown or Not Reported | 3 | 2 | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian/Alaskan Native | 6 | 8 | 14
  Asian | 8 | 5 | 13
  Black/African American | 22 | 23 | 45
  White/Caucasian | 197 | 201 | 398
  Native Hawaiian/Pacific Islander | 4 | 5 | 9
  South Asian | 3 | 2 | 5
  Unknown/Not reported | 17 | 22 | 39
  Other (identified as other) | 29 | 21 | 50
SPO2 [Mean (Standard Deviation); unit: mmHg] — This is a scale measuring your level of oxygen. A level of 95% or more is considered normal.
  mmHg | 96.8 (12.7) | 96.8 (13.5) | 96.8 (1.7)
Duration of Covid-19 symptoms [Mean (Standard Deviation); unit: days] — How many days COVID-19 symptoms lasted at baseline.This would mean the number of days since the onset of symptoms at the time the participant enrolled.
  days | 5 (1.44) | 4.8 (1.52) | 4.9 (1.49)
Coexisting conditions [Count of Participants; unit: Participants]
  Heart disease | 4 | 4 | 8
  Lung disease | 2 | 2 | 4
  Liver disease | 1 | 1 | 2
  Kidney disease | 1 | 2 | 3
  Hepatitis B/C | 1 | 1 | 2
  Immune disorder | 14 | 4 | 18
  HIV | 1 | 4 | 5
  Asthma | 40 | 33 | 73
  Hypertension | 55 | 62 | 117
  Diabetes | 23 | 28 | 51
  Active cancer | 0 | 1 | 1
  Thyroid problem | 20 | 27 | 47
  Other medical conditions | 42 | 54 | 96
Most severe COVID-19 symptom at baseline [Count of Participants; unit: Participants] — Some people reported more than one symptom as their most severe symptom. This means some of the participants can be represented in more than one row.
  Participants
    Loss of smell | 74 | 91 | 165
    Fatigue | 70 | 59 | 129
    Loss of taste | 47 | 48 | 95
    Nasal congestion | 45 | 30 | 75
    Cough | 34 | 37 | 71
    Body aches | 27 | 30 | 57
    Loss of appetite | 21 | 26 | 47
    Subjective fever | 12 | 18 | 30
    Nausea | 11 | 4 | 15
    Chills | 9 | 10 | 19
    Diarrhea | 8 | 9 | 17
    Sore throat | 8 | 7 | 15
    Shortness of breath | 6 | 7 | 13
Body Mass Index category (BMI) [Count of Participants; unit: Participants] — A BMI measurement of 25 and under means normal to underweight range. A measurement of 25-29.9 means overweight range. Measurements of 30 and over mean obese range.
  Participants
    Less than 25 | 71 | 62 | 133
    25-29.9 | 86 | 90 | 176
    Greater than or equal to 30 | 115 | 123 | 238

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Clinical Deterioration
Description: Defined as the number of participants who experienced the following: both of the following: 1)Presence of dyspnea and/or hospitalization for shortness of breath or pneumonia, 2)) decrease in O2 saturation (<92% on room air) and/or supplemental oxygen requirement to keep O2 saturation ≥92%).
Time Frame: RCT-approximately 15 days
Measure: Count of Participants; unit: Participants
Arm/Group | Fluvoxamine | Placebo
Number analyzed (Participants) | 272 | 275
Participants | 13 | 15

ADVERSE EVENTS:
Time Frame: Approximately 90 days
Arm/Group | Fluvoxamine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/272 | 0/275
Serious Adverse Events (participants affected / at risk) | 13/272 | 12/275
Other Adverse Events (participants affected / at risk) | 15/272 | 5/275
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fluvoxamine (N=272) | Placebo (N=275)
Appendicitis (General disorders) | 0 (0) | 1 (1)
Bowel issues (General disorders) | 1 (1) | 0 (0) — one instance of bowel blockage requiring hospitalization
Dry mouth (General disorders) | 1 (1) | 1 (1)
Breathing problems (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 5 (5) — including shortness of breath, and low oxygen
Pneumonia (Infections and infestations) | 6 (6) | 1 (1)
Pulmonary embolism (General disorders) | 0 (0) | 1 (1)
Skin reaction (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — one instance of staphylococcal skin/soft tissue infection of upper extremity requiring hospitalization.
Vertigo (General disorders) | 0 (0) | 1 (1) — vertigo/vision problems
Worsening of COVID symptoms (Infections and infestations) | 1 (1) | 2 (2) — requiring hospitalization
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fluvoxamine (N=272) | Placebo (N=275)
Nausea/vomitting (General disorders) | 15 (15) | 5 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-04-14): https://cdn.clinicaltrials.gov/large-docs/50/NCT04668950/Prot_000.pdf
  • Statistical Analysis Plan (2021-11-15): https://cdn.clinicaltrials.gov/large-docs/50/NCT04668950/SAP_001.pdf